CLINICAL TRIAL: NCT03953716
Title: Clinical and Systematic Biology Study of Traditional Chinese Medicine, Western Medicine and Low-level Light Therapy for Primary
Brief Title: Traditional Chinese Medicine, Western Medicine and Low-level Light Therapy（LLLT） for Primary Dysmenorrhea（PD）
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Aijun Sun, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PD201903
Record Dates: First submitted 2019-04-14; First posted 2019-05-17 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Primary Dysmenorrhea; Traditional Chinese Medicine; Light
Keywords: Primary Dysmenorrhea; traditional Chinese medicine; low-level light therapy
MeSH Terms: interventions — Low-Level Light Therapy; Desogestrel

STUDY DESIGN:
Intervention Model Description: One fourth of participants will receive Ding Kun Dan Pills, one fourth of participants will receive Simulated drug of DING KUN DAN Pills, one fourth of participants will receive MARVELON ,and the another fourth will receive low level light therapy
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DING KUN DAN (Experimental): DING KUN DAN,3.5g BID for 10 days (starting 3-5 days before menstruation) *3 menstrual cycle
  Interventions: Drug: DING KUN DAN
- Simulated drug of DING KUN DAN (Placebo Comparator): Simulated drug of DING KUN DAN，3.5g BID for 10 days (starting 3-5 days before menstruation) *3 menstrual cycle
  Interventions: Drug: Simulated drug of DING KUN DAN
- low level light therapy (Experimental): Start using low level light therapy after the menstrual period, once a day, every 20 minutes * 5 days ( one treatment cycle), start the next course at intervals of 2 days until the next menstruation
  Interventions: Device: low level light therapy
- Marvelon (Active Comparator): 1 pill QD*21 days (starting on the 5th day of menstruation, continuing the next cycle after 1 week of withdrawal) *3 menstrual cycle
  Interventions: Drug: Marvelon

INTERVENTIONS:
Device: low level light therapy — Start using low level light therapy after the menstrual period, once a day, every 20 minutes * 5 days ( one treatment cycle), start the next course at intervals of 2 days until the next menstruation
  Arms: low level light therapy
Drug: DING KUN DAN — DING KUN DAN,3.5g BID for 10 days (starting 3-5 days before menstruation) *3 menstrual cycle
  Arms: DING KUN DAN
Drug: Simulated drug of DING KUN DAN — Simulated drug of DING KUN DAN，3.5g BID for 10 days (starting 3-5 days before menstruation) *3 menstrual cycle
  Arms: Simulated drug of DING KUN DAN
Drug: Marvelon — Marvelon 1 pill QD*21 days (starting on the 5th day of menstruation, continuing the next cycle after 1 week of withdrawal) *3 menstrual cycle
  Arms: Marvelon

SUMMARY:
To observe the clinical efficacy and safety of three methods for the treatment of primary dysmenorrhea. Establish an integrated biomarker index system for the evaluation of the efficacy of traditional Chinese medicine, western medicine and Low-level Light Therapy for the treatment of primary dysmenorrhea, and further explore the mechanism and therapeutic material basis of the three treatment methods for the treatment of primary dysmenorrhea

DETAILED DESCRIPTION:
480 women clinically diagnosed of primary dysmenorrhea will be enrolled from nationwide multi-centers. Blood samples were collected from 480 patients before and after treatment (1 experimental group, 3 control groups, treatment cycle of 3 menstrual cycles, follow-up cycle of 5 menstrual cycles), Metabonomics study, and integration of clinical sample information (Serum biochemical indicators, imaging indicators, etc.), through bioinformatics to establish a comprehensive biomarker index system for the evaluation of the efficacy of traditional Chinese medicine, Western medicine and Low-level Light Therapy instrument Methods for the treatment of primary dysmenorrhea and its therapeutic basis.

ELIGIBILITY:
Inclusion Criteria:

1. Female (16-35 years old);
2. regular Menstruation (cycle 21-35 days, menstrual period 3-7 days);
3. Be clinically diagnosed with primary dysmenorrhea;
4. Be willing to participate in the whole process of the research in 5 consecutive menstrual cycles.

Exclusion Criteria:

1. irregular menstruation affecting the treatment and efficacy judgment;
2. Patients with secondary dysmenorrhea;
3. Those who have used related drugs in the past 3 months;
4. Abuse or dependence on substances (alcohol or medicine) in the past 3 months; heavy smokers (smokers who smoke 20 or more cigarettes per day);
5. Those who have severe or unstable physical illnesses, related to liver, kidney, gastrointestinal tract, cardiovascular, respiratory, endocrine, nervous, immune or blood systems, neuropsychiatric systems and so on;
6. Lactating or pregnant women, or women within 1 year after delivery;
7. Those who are allergic to the test drug or light, have contraindications for Marvelon and Ding kun dan;
8. Have a history of thromboembolic disease or a tendency to thrombosis;
9. one month before joining in this study (first interview), Who participated in another clinical trial;
10. Those who meet the inclusion criteria, fail to follow the doctor's advice so that we cannot judge the curative effect ,the incomplete data cannot be evaluated.

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 480 (Estimated)
Dates: Start 2019-06-22 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale,VAS | about 30 days
  Visual Analogue Scale/Score (VAS): Draw a 10 cm horizontal line on the paper. The degree of pain is indicated by the line segment，One end of the horizontal line is 0, indicating no pain; the other end is 10, indicating severe pain; the middle part indicates different degrees of pain（the mild pain is 1-3, the moderate is 4-6, the severity is 7-9），The patient chooses the value that can represent the degree of pain.

SECONDARY OUTCOMES:
Short-form McGill Pain Questionnaire-2, SF-MPQ-2 | about 30 days
  Short-form McGill Pain Questionnaire-2(SF-MPQ-2), By this scale, we can evaluate the different types of pain and the emotional effects of PD. It has 22 entries. These 22 entries include: Jumping pain, shooting pain, knife-like pain, sharp pain, cramping and dragging pain, constant biting pain, hot burning pain, sore pain, falling pain, slightly pressing pain, tearing pain, exhaustion - weakness, disgusting, fear, Torture - punishment, electric shock, cold pain, puncture pain, pain caused by gentle touch, itching, pin and needles pain, numbness. Each entry scored "0~10" points, the minimum score is 0,the maximum score is 10,a total of 11 levels. "0" indicates that never have this pain or symptom, "10" represents that this pain or feel is severe,"1-9" indicates different degrees of this type of pain or symptom. At last, Calculate the total score of all 22 items.
the COX menstrual symptom scale，CMSS | about 30 days
  the COX menstrual symptom scale (CMSS), this score evaluate the level of PD from the two aspects of dysmenorrhea symptoms: the duration and severity , It has 17 entries including: cramps , nausea, vomiting, loss of appetite, headaches, backaches, leg aches, dizziness, weakness, diarrhea, facial blemishes, abdominal pain, flushing, general aching, depression, irritability, nervousness. Each entry scored "0~4" points, different score represents different duration or severity of corresponding symptoms : for the duration, 0 indicates never have this symptom, 1 means lasting less 3 hours, 2 means lasting 3~7 hours, 3 means 7~24 hours, 4 means more than 24 hours. as for the severity,0 indicates no pain; the mild is 1, the moderate is 2, the severity is 3, the extreme severity is 4. Then, Calculate the score of the duration and severity of all 17 items respectively, lastly, sum the total score of the duration and severity.
Menstrual flow graph analysis table | about 30 days
  Through this form, we can know about the menstrual period and menstrual flow before and after treatment:
  Mild: blood stained area ≤ 1/3 of the entire sanitary napkin area; Moderate: blood stained area accounts for 1/3-3/5 of the entire sanitary napkin area; Severe: The blood stained area is basically the entire sanitary napkin. Blood clot area <1 dollar coin, which is a small blood clot; The blood clot area is ≥1 yuan coin, which is a large blood clot. fill in the number of sanitary napkins used in the appropriate space according to the degree of blood stain or the amount of the blood clot on each sanitary napkin discarded.
Uterine artery Pulsation index | 3 months
  Determination of uterine artery hemodynamics, can reflect the state of uterine blood circulation, the higher the uterine artery pulsation index, the decrease of blood flow, the lower the uterine artery pulsation index, the increase of blood flow or neo-vascularization
Uterine artery Resistance index | 3 months
  Determination of uterine artery hemodynamics, can reflect the state of uterine blood circulation, the higher the uterine artery resistance index, indicating less blood supply to uterine, the lower the uterine artery resistance index, the increased blood supply to uterine.
Uterine artery Systolic peak and diastolic peak ratio | 3 months
  The greater the ratio of uterine artery systolic peak to diastolic peak, indicating that the end-diastolic blood flow velocity is small and the peripheral resistance is large; conversely, the blood flow velocity is large and the peripheral resistance is small.

CONTACTS AND LOCATIONS:
Overall Officials: Aijun SUN, MD, Principal Investigator — Peking Union Medical College Hospital, Chinese Academy of Medicine Sciences
Locations (1):
- Xiao MA, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Network platform, and the website will be attached later.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Within six months after the trial complete
Access Criteria: Data access requests will be reviewed by an external independent review panel.Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Zhu S, Ma X, Ding X, Gan J, Deng Y, Wang Y, Sun A. Comparative evaluation of low-level light therapy and ethinyl estradiol and desogestrel combined oral contraceptive for clinical efficacy and regulation of serum biochemical parameters in primary dysmenorrhoea: a prospective randomised multicentre trial. Lasers Med Sci. 2022 Jun;37(4):2239-2248. doi: 10.1007/s10103-021-03490-z. Epub 2022 Jan 14. PMID 35028764